CLINICAL TRIAL: NCT02106663
Title: Evaluating the Efficacy of Circumferential Pulmonary Vein Ablation (CPVA) Versus Segmental Pulmonary Vein Isolation (SPVI) in Paroxysmal Atrial Fibrillation
Brief Title: Effectiveness Study of Circumferential vs. Segmental Ablation in Paroxysmal Atrial Fibrillation
Acronym: PAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Greg Feld, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110531
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Paroxysmal Atrial Fibrillation; Atrial Arrhythmia
Keywords: atrial fibrillation; paroxysmal atrial fibrillation; PAF; arrhythmia; atrial fibrillation ablation; circumferential ablation; CPVA; segmental ablation; PVI; pulmonary vein isolation
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Circumferential Pulmonary Vein Ablation (Active Comparator): Contiguous ablation lesions will be performed to encircle the two left and right pulmonary veins (PVs), guided by 3D electroanatomic mapping (Carto, Biosense Webster, Inc. or ESI NavX, St. Jude, Inc.) with a 3D LA geometry created either by using the roving mapping catheter or by importing a pre-recorded 3D CT image of the left atrium. After completion of the circumferential ablation, PV isolation will be confirmed by the mapping catheter, and further focal ablation performed as required until electrical PV isolation is confirmed (entrance block at a minimum).
  Interventions: Procedure: Circumferential Pulmonary Vein Ablation
- Segmental Pulmonary Vein Isolation (Active Comparator): Electrical potentials recorded in the pulmonary vein (PV) ostium using a circular mapping catheter, representing myocardial connections between the left atrium and PVs will be ablated at or just proximal to the PV ostium in the PV antrum. Ablation will be performed segmentally at multiple sites guided by the mapping catheter around the PV ostium or antrum, until mapping demonstrates elimination of all PV potentials (entrance block at a minimum).
  Interventions: Procedure: Segmental Pulmonary Vein Isolation

INTERVENTIONS:
Procedure: Circumferential Pulmonary Vein Ablation — Contiguous ablation lesions will be performed to encircle the two left and right pulmonary veins (PVs) of the left atrium, guided by 3D electroanatomic mapping. After completion of the circumferential ablation, PV isolation will be confirmed by the mapping catheter, and further focal ablation performed as required until electrical PV isolation is confirmed.
  Other Names: radiofrequency catheter ablation; atrial fibrillation ablation
  Arms: Circumferential Pulmonary Vein Ablation
Procedure: Segmental Pulmonary Vein Isolation — Electrical potentials recorded in the pulmonary vein (PV) ostium using a circular mapping catheter, representing electrical connections between the left atrium and PVs will be ablated at or just proximal to the PV ostium in the PV antrum. Ablation will be performed segmentally at multiple sites guided by the mapping catheter until mapping demonstrates elimination of all PV potentials.
  Other Names: radiofrequency catheter ablation; atrial fibrillation ablation
  Arms: Segmental Pulmonary Vein Isolation

SUMMARY:
This is a PI-initiated study that aims to evaluate the efficacy of two different methods of paroxysmal atrial fibrillation (PAF) ablation. There are currently two strategies for PAF ablation that are routinely performed by electrophysiology clinicians: (1) circumferential pulmonary vein ablation (CPVA) and (2) segmental pulmonary vein isolation (SPVI). However, it is not known if one approach is better than the other. This randomized study will evaluate and compare the efficacy of CPVA versus SPVI in subjects undergoing ablation for paroxysmal atrial fibrillation only. Subjects will have a 50/50 chance of receiving either the CPVA or SPVI ablation method.

DETAILED DESCRIPTION:
Despite more than a decade of clinical experience and investigation, the optimal approach to ablation of paroxysmal atrial fibrillation (PAF) still remains controversial. There are currently two strategies for ablation of PAF: (1) circumferential pulmonary vein ablation (CPVA) and (2) segmental pulmonary vein isolation (SPVI). There are advantages and disadvantages associated with each method. In the CPVA method (1), contiguous ablation lesions are created to encircle the two left and right pulmonary veins (PVs), guided by a three-dimensional (3D) electroanatomic mapping system (Carto, Biosense Webster, Inc. or ESI NavX, St. Jude, Inc.) with a 3D left atrial (LA) geometry created either by using the mapping catheter or by importing a pre-recorded 3D computed tomography (CT) image. In the SPVI method (2), electrical potentials recorded at the PV ostium, that represent myocardial connections between the LA and PVs, are ablated at the PV ostium or just proximal to the PV ostium in the PV antrum. In this approach, ablation is performed segmentally at multiple sites around the PV ostium or antrum, until mapping with a circular catheter demonstrates pulmonary vein isolation.

The reported success rates for SPVI for prevention of recurrence of PAF range from 60-87% (2-4) with most recurrences associated with recovery of PV conduction. Therefore, the success of SPVI for treatment of PAF appears to be related to in large part to permanent elimination of the triggers of AF. In a retrospective study by Sawhney et al, overall 5-year outcome after SPVI for PAF was similar to that for short-term follow up less than or equal to 2 years. However, late recurrences after 2 years did occur (up to 22.5%) and repeat ablation was often required to maintain freedom from symptomatic PAF (5).

Even though success rates for CPVA have been reported to be higher (up to 90%), most CPVA procedures previously reported included left atrial linear ablation (LALA), additional ablation lesions or lines connecting the mitral valve to the posterior pulmonary veins or along the roof of the left atrium. Thus the success of CPVA may be due in part to ablation of substantially larger amounts of atrial tissue (6-7). However, additional ablation (LALA) may cause potential pro-arrhythmic effects that lead to development of atypical left atrial flutter (8).

Compared to SPVI, CPVA resulted in higher success rates and lower fluoroscopy time in one study by Arentz et al (9). However, that study included subjects with both PAF and persistent AF, and those with persistent AF have potentially different underlying mechanisms. Furthermore, two other randomized studies comparing the efficacy of PVI and CPVA have shown conflicting results (10-11).

Thus, we will initiate this randomized controlled study to evaluate the efficacy of CPVA versus SPVI in subjects undergoing ablation of paroxysmal atrial fibrillation only.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with paroxysmal atrial fibrillation, whose episodes have never been documented to exceed 48 hours duration
2. Patients with a clinical indication for ablation
3. Patients greater than 18 years of age.
4. Patients willing and able to give informed consent.
5. Patients with concurrent atrial fibrillation and atrial flutter are allowed.

Exclusion Criteria:

1. Patients with medical conditions that would limit participation for the entire duration of the study.
2. Patients that are pregnant (all females of child-bearing potential must have a negative pregnancy test within 1 week of enrollment).
3. Patients having undergone prior AF ablation
4. Patients with paroxysmal atrial fibrillation whose episodes last greater than 48 hours
5. Patients with persistent AF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Atrial Fibrillation Recurrence | 2 years
  Recurrence of atrial fibrillation (AF) will be defined as any ECG documented symptomatic AF, or asymptomatic AF lasting >30 seconds on Mobile Outpatient Cardiac Telemetry (MCOT) monitoring. Subjects will be scheduled for clinic visits at 1, 6, 12 and 24 months post ablation. In addition, mobile outpatient telemetry will be performed for at least seven days at 6, 12 and 24 months post-procedure to detect recurrence of asymptomatic atrial fibrillation.

SECONDARY OUTCOMES:
Pulmonary Vein Stenosis | 3 Months
  A CT scan of the left atrium and pulmonary veins will be routinely performed 3 months after ablation to assess for any evidence of pulmonary vein stenosis

CONTACTS AND LOCATIONS:
Overall Officials: Gregory K Feld, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Sulpizio Cardiovascular Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feld GK, Sawhney N. What is the optimal approach for ablation of paroxysmal atrial fibrillation? Heart Rhythm. 2009 Aug;6(8 Suppl):S23-8. doi: 10.1016/j.hrthm.2009.03.002. Epub 2009 Mar 3. PMID 19410519
- [Background] Shah DC, Haissaguerre M, Jais P, Hocini M, Yamane T, Deisenhofer I, Garrigue S, Clementy J. Electrophysiologically guided ablation of the pulmonary veins for the curative treatment of atrial fibrillation. Ann Med. 2000 Sep;32(6):408-16. doi: 10.3109/07853890008995948. PMID 11028689
- [Background] Oral H, Knight BP, Tada H, Ozaydin M, Chugh A, Hassan S, Scharf C, Lai SW, Greenstein R, Pelosi F Jr, Strickberger SA, Morady F. Pulmonary vein isolation for paroxysmal and persistent atrial fibrillation. Circulation. 2002 Mar 5;105(9):1077-81. doi: 10.1161/hc0902.104712. PMID 11877358
- [Background] Oral H, Knight BP, Ozaydin M, Chugh A, Lai SW, Scharf C, Hassan S, Greenstein R, Han JD, Pelosi F Jr, Strickberger SA, Morady F. Segmental ostial ablation to isolate the pulmonary veins during atrial fibrillation: feasibility and mechanistic insights. Circulation. 2002 Sep 3;106(10):1256-62. doi: 10.1161/01.cir.0000027821.55835.00. PMID 12208802
- [Background] Sawhney N, Anousheh R, Chen WC, Narayan S, Feld GK. Five-year outcomes after segmental pulmonary vein isolation for paroxysmal atrial fibrillation. Am J Cardiol. 2009 Aug 1;104(3):366-72. doi: 10.1016/j.amjcard.2009.03.044. Epub 2009 Jun 6. PMID 19616669
- [Background] Pappone C, Rosanio S, Oreto G, Tocchi M, Gugliotta F, Vicedomini G, Salvati A, Dicandia C, Mazzone P, Santinelli V, Gulletta S, Chierchia S. Circumferential radiofrequency ablation of pulmonary vein ostia: A new anatomic approach for curing atrial fibrillation. Circulation. 2000 Nov 21;102(21):2619-28. doi: 10.1161/01.cir.102.21.2619. PMID 11085966
- [Background] Pappone C, Oreto G, Rosanio S, Vicedomini G, Tocchi M, Gugliotta F, Salvati A, Dicandia C, Calabro MP, Mazzone P, Ficarra E, Di Gioia C, Gulletta S, Nardi S, Santinelli V, Benussi S, Alfieri O. Atrial electroanatomic remodeling after circumferential radiofrequency pulmonary vein ablation: efficacy of an anatomic approach in a large cohort of patients with atrial fibrillation. Circulation. 2001 Nov 20;104(21):2539-44. doi: 10.1161/hc4601.098517. PMID 11714647
- [Background] Sawhney N, Anousheh R, Chen W, Feld GK. Circumferential pulmonary vein ablation with additional linear ablation results in an increased incidence of left atrial flutter compared with segmental pulmonary vein isolation as an initial approach to ablation of paroxysmal atrial fibrillation. Circ Arrhythm Electrophysiol. 2010 Jun;3(3):243-8. doi: 10.1161/CIRCEP.109.924878. Epub 2010 Mar 25. PMID 20339034
- [Background] Arentz T, Weber R, Burkle G, Herrera C, Blum T, Stockinger J, Minners J, Neumann FJ, Kalusche D. Small or large isolation areas around the pulmonary veins for the treatment of atrial fibrillation? Results from a prospective randomized study. Circulation. 2007 Jun 19;115(24):3057-63. doi: 10.1161/CIRCULATIONAHA.107.690578. Epub 2007 Jun 11. PMID 17562956
- [Background] Oral H, Scharf C, Chugh A, Hall B, Cheung P, Good E, Veerareddy S, Pelosi F Jr, Morady F. Catheter ablation for paroxysmal atrial fibrillation: segmental pulmonary vein ostial ablation versus left atrial ablation. Circulation. 2003 Nov 11;108(19):2355-60. doi: 10.1161/01.CIR.0000095796.45180.88. Epub 2003 Oct 13. PMID 14557355
- [Background] Karch MR, Zrenner B, Deisenhofer I, Schreieck J, Ndrepepa G, Dong J, Lamprecht K, Barthel P, Luciani E, Schomig A, Schmitt C. Freedom from atrial tachyarrhythmias after catheter ablation of atrial fibrillation: a randomized comparison between 2 current ablation strategies. Circulation. 2005 Jun 7;111(22):2875-80. doi: 10.1161/CIRCULATIONAHA.104.491530. Epub 2005 May 31. PMID 15927974
- [Background] Calkins H, Kuck KH, Cappato R, Brugada J, Camm AJ, Chen SA, Crijns HJ, Damiano RJ Jr, Davies DW, DiMarco J, Edgerton J, Ellenbogen K, Ezekowitz MD, Haines DE, Haissaguerre M, Hindricks G, Iesaka Y, Jackman W, Jalife J, Jais P, Kalman J, Keane D, Kim YH, Kirchhof P, Klein G, Kottkamp H, Kumagai K, Lindsay BD, Mansour M, Marchlinski FE, McCarthy PM, Mont JL, Morady F, Nademanee K, Nakagawa H, Natale A, Nattel S, Packer DL, Pappone C, Prystowsky E, Raviele A, Reddy V, Ruskin JN, Shemin RJ, Tsao HM, Wilber D; Heart Rhythm Society Task Force on Catheter and Surgical Ablation of Atrial Fibrillation. 2012 HRS/EHRA/ECAS expert consensus statement on catheter and surgical ablation of atrial fibrillation: recommendations for patient selection, procedural techniques, patient management and follow-up, definitions, endpoints, and research trial design: a report of the Heart Rhythm Society (HRS) Task Force on Catheter and Surgical Ablation of Atrial Fibrillation. Developed in partnership with the European Heart Rhythm Association (EHRA), a registered branch of the European Society of Cardiology (ESC) and the European Cardiac Arrhythmia Society (ECAS); and in collaboration with the American College of Cardiology (ACC), American Heart Association (AHA), the Asia Pacific Heart Rhythm Society (APHRS), and the Society of Thoracic Surgeons (STS). Endorsed by the governing bodies of the American College of Cardiology Foundation, the American Heart Association, the European Cardiac Arrhythmia Society, the European Heart Rhythm Association, the Society of Thoracic Surgeons, the Asia Pacific Heart Rhythm Society, and the Heart Rhythm Society. Heart Rhythm. 2012 Apr;9(4):632-696.e21. doi: 10.1016/j.hrthm.2011.12.016. Epub 2012 Mar 1. No abstract available. PMID 22386883
- [Background] Wann LS, Curtis AB, January CT, Ellenbogen KA, Lowe JE, Estes NA 3rd, Page RL, Ezekowitz MD, Slotwiner DJ, Jackman WM, Stevenson WG, Tracy CM; 2006 WRITING COMMITTEE MEMBERS; Fuster V, Ryden LE, Cannom DS, Le Heuzey JY, Crijns HJ, Lowe JE, Curtis AB, Olsson S, Ellenbogen KA, Prystowsky EN, Halperin JL, Tamargo JL, Kay GN, Wann LS; ACCF/AHA TASK FORCE MEMBERS; Jacobs AK, Anderson JL, Albert N, Hochman JS, Buller CE, Kushner FG, Creager MA, Ohman EM, Ettinger SM, Stevenson WG, Guyton RA, Tarkington LG, Halperin JL, Yancy CW. 2011 ACCF/AHA/HRS focused update on the management of patients with atrial fibrillation (Updating the 2006 Guideline): a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Heart Rhythm. 2011 Jan;8(1):157-76. doi: 10.1016/j.hrthm.2010.11.047. Epub 2010 Dec 21. No abstract available. PMID 21182985